CLINICAL TRIAL: NCT00273130
Title: Randomised Evaluation of Neuroendocrine Stress Response During Upper Gastrointestinal Endoscopy With Standard or Ultrathin Endoscope.
Brief Title: Stress Response Using Thin and Standard Size Endoscopy.
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MC-01-KAT; KF01-245/97
Record Dates: First submitted 2006-01-05; First posted 2006-01-09 (Estimated); Last update posted 2006-09-13 (Estimated); Status verified 2003-12

CONDITIONS: Upper Gastrointestinal Disease,Ulcers
Keywords: transnasal gastroscopy, stress response, ischaemia
MeSH Terms: conditions — Gastrointestinal Diseases; Ulcer; Fractures, Stress; Ischemia

INTERVENTIONS:
Procedure: transnasal endoscopy
Procedure: transoral thin endoscopy

SUMMARY:
Sixty patients scheduled for upper diagnostic gastroscopy were randomised after written informed consent into three groups.

1. transnasal gastroscopy with thin endoscope
2. transoral with thin endoscope
3. standard size trans-oral endoscopy Stress response parameters (epinephrine, nor-epinephrine and cortisol, heartrate variability data and pulse oximetry data were monitored.

DETAILED DESCRIPTION:
A substantial number of descriptive studies and clinical trials have made it evident that upper gastrointestinal endoscopy elicits cardiovascular and respiratory changes. Recent publications have indicated less marked cardiovascular changes when using thinner endoscopes or transnasal endoscopy .Hormonal stress response during upper gastrointestinal endoscopy has also been described, but never related to the different methods of upper gastrointestinal endoscopy. Furthermore the patient tolerance is markedly improved compared to the standard transoral route.

The aim of the present randomised study was to evaluate the ECG-, blood pressure- and pulse rate changes and the endocrine stress response (norepinephrine, epinephrine and cortisol) elicited by upper gastrointestinal endoscopy using a thin endoscope either transnasally or orally or a standard endoscope orally.

Method and material Sixty patients were included consecutively after written and informed consent and were all over 18 years. Patients receiving digitalis, ß-blocking agents or calcium antagonists were excluded, as well as patients receiving drugs for thyroid dysfunction or patients receiving steroids. Patients with known disease or trauma of the nasal cavity were not included.

Only intended diagnostic upper gastrointestinal endoscopies were included. The patients received standard medication during the endoscopy if required.

Immediately prior to the endoscopy each of the 60 patients chose an envelope with the allocation to one of three groups A) Endoscopy with a thin endoscope (4.5 mm Olympus prototype fiberendoscope) introduced transnasally (T group), B) Endoscopy with a thin endoscope (4.5 mm Olympus prototype fiberendoscope) introduced orally (O group) or C) Endoscopy with a standard gastroscope (6 mm Olympus GIF XV10) (S group). All patients received the same amount of a local anesthetic spray (Lidocaine 10 mg/dose, ASTRA Zeneca) (twice in each nostril and twice in the oropharynx, given by one of two particular persons to ensure application of comparable doses of local anesthetic).

ELIGIBILITY:
Inclusion Criteria:

* diagnostic gastroscopy, age over 18, danish speaking,

Exclusion Criteria:

* use of beta blocking or any other heart rate modulating drug, antithyroid drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 1999-03; Study Completion 2002-08

PRIMARY OUTCOMES:
tachycardia, ischaemia, level of stress response

SECONDARY OUTCOMES:
acceptability of transnasal endoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Merete Christensen, MD, Principal Investigator — Dept of Cardiothoracic Surgery, Copenhagen University Hospital, Rigshospitalet, Copenhagen
Locations (1):
- Hvidovre University Hospital, Dept of Surgery, Hvidovre, Denmark